CLINICAL TRIAL: NCT05523960
Title: Mechanical Bowel Preparation Versus no Bowel Preparation for Esophageal Cancer Surgery: a Multi-center, Randomized, Parallel, Single-blinded Trial
Brief Title: Mechanical Bowel Preparation Versus no Bowel Preparation for Esophageal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCC2020C-511
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBP group (Experimental): Patients allocated to NBP were instructed to not prepare the bowel.
  Interventions: Procedure: No MBP
- MBP group (Other): Patients allocated to MBP were instructed by the study nurse to prepare their bowel mechanically by drinking 3~4L of polyethylene glycol (Polyethylene Glycol Electrolytes Powder 68.56g; Shenzhen, China) with water before 6pm in the evening the day before the surgery.
  Interventions: Procedure: No MBP

INTERVENTIONS:
Procedure: No MBP — No mechanical bowel preparation before operation

SUMMARY:
The study type was designed as a prospective multicenter randomized controlled study. The patients will be divided into intervention group and control group, 281 patients were needed for each group and 562 patients would be needed totally to show this difference. Due to a possible loss of 14%, the final sample size was calculated to be 652 patients. The intervention group will not implement mechanical bowel preparation(MBP) before surgery; the control group will receive routine preoperative MBP for oral administration of compound polyethylene glycol electrolyte powder and fasting water. Perioperative complications, intestinal recovery speed and quality of life will be investigated between the two groups.

DETAILED DESCRIPTION:
Patients allocated to MBP will be instructed by the study nurse to prepare their bowel mechanically by drinking 3~4L of polyethylene glycol (Polyethylene Glycol Electrolytes Powder 68.56g; Shenzhen, China) with water before 6pm in the evening the day before the surgery. Patients allocated to NBP were instructed to not prepare the bowel. The receipt of the allocated intervention will be controlled by study nurse asking the patients on the morning of the surgery whether they had acted as instructed by the allocation. This information will be also concealed from treating physicians and surgeons, data collectors, and data analysts, until the primary and secondary outcomes were analyzed. All patients will follow the ERAS protocol. Prophylactic intravenous antibiotics (cephamycin 1000mg) will be given to all patients 30 minutes before skin incision. The prophylactic intravenous antibiotics will re-administered if the surgery lasted longer than 3h from the first antibiotic dose. Surgical skin preparation will involve taking a bath well the night before operation without shaving the hair. Just before skin incision, the area will then washed three times with denatured 80% alcohol to left to dry.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were scheduled for esophageal cancer resection in participating centers were eligible for inclusion.

Exclusion Criteria:

* need for emergency surgery;
* previous chronic constipation or diarrhea;
* previous abdominal surgery; need for colonic reconstruction;
* other indications for mechanical preparation or contraindications;
* allergy to drugs used in the trial (polyethylene glycol)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
the rate of major complications | during surgery orwithin 30 days after surgery
  A major intraoperative and postoperative complication was defined as a surgical or medical complication with a Clavien-Dindo (CD) grade of Ⅱor higher (this five-grade system includes sub-grades in grades Ⅲ and Ⅳ, and higher grades indicate more life-threatening complications) according to Esophagectomy Complications Consensus Group (ECCG)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No